CLINICAL TRIAL: NCT02804919
Title: CPAP In-home Assessment NZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA174
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational CPAP device (Experimental): Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: Fisher & Paykel Healthcare CPAP Device

INTERVENTIONS:
Device: Fisher & Paykel Healthcare CPAP Device — Fisher & Paykel Healthcare CPAP Device

SUMMARY:
Phase 1:The study is to evaluate the product reliability, therapy effectiveness and user feedback of a Continuous Positive Airway Pressure (CPAP) device in-home for up to 6 months.

Phase 2: To evaluate the CPAP device with communication functionality with data upload.

DETAILED DESCRIPTION:
Phase 1:Existing and Naïve CPAP users will be recruited into a 6 month in-home study Participants will attend 5 study visits at day 0, 7, 30, 60 and 180. Outcome of the clinical investigation include downloadable device data reports, device error reports and participants perception questionnaires.

Phase 2: 10 participants from Phase 1 will be recruited to use the device for up to 6 month in-home. Participants will attend 3 study visits at day 0, 7 30. The trial may be extended to 60 days if longer term data is required.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Diagnosed with Obstructive Sleep Apnea (OSA) and prescribed Positive Airway Pressure (either Continuous positive airway pressure (CPAP) or AutoCPAP)
* Be fluent in spoken and written English

Exclusion Criteria:

* Contraindicated for Positive Airway Pressure (CPAP or AutoCPAP) therapy
* Persons with other significant sleep disorder(s) (e.g periodic leg movements, insomnia, central sleep apnea)
* Persons with obesity hypoventilation syndrome or congestive heart failure
* Persons that require supplemental oxygen with their Positive Airway Pressure (CPAP or AutoCPAP) device.
* Persons with implanted electronic medical devices (e.g cardiac pacemakers)
* Persons who are pregnant or think they may be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI), measured as number of events/hour hour. | 6 months
  Obtained from the device - Phase 1 and Phase 2 of the trial
Log of safety-related events, measured as number of safety-related faults | 6 months
  Obtained from the device - Phase 1 and Phase 2 of the trial
Machine reported faults, measured as number of machine faults | 6 months
  Obtained from the device - Phase 1 and Phase 2 of the trial
Participant reported faults, measured as number of participant complaints | 6 months
  Obtained from the follow up visits - Phase 1 and Phase 2 of the trial

SECONDARY OUTCOMES:
Perception of the device, measured through questionnaire | 6 months
  Impression of the device during the follow up visits - Phase 1 only

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cheung, MSc/RPSGT, Principal Investigator — Fisher & Paykel Healthcare
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand